CLINICAL TRIAL: NCT02812472
Title: Treadmill Training With Functional Electric Stimulation in Patients With Chronic Stroke
Brief Title: Treadmill Training With Functional Electric Stimulation After Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 960053
Record Dates: First submitted 2016-06-15; First posted 2016-06-24 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-06

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

ARMS (2):
- treadmill training with functional electrical stimulation (Experimental): Subjects in the experimental group received additional treadmill training with functional electric stimulation for 25 minutes per session, followed by 5 minutes cool down for 12 sessions.
  Interventions: Other: Treadmill training with functional electrical stimulation
- treadmill training without functional electrical stimulation (Active Comparator): Subjects in the control group received additional treadmill training without functional electric stimulation for 25 minutes per session, followed by 5 minutes cool down for 12 sessions.
  Interventions: Other: Treadmill training without functional electrical stimulation

INTERVENTIONS:
Other: Treadmill training with functional electrical stimulation
  Arms: treadmill training with functional electrical stimulation
Other: Treadmill training without functional electrical stimulation
  Arms: treadmill training without functional electrical stimulation

SUMMARY:
The purpose of this study was to investigate the effects of the treadmill training with functional electric stimulation on sensorimotor cortical reorganization and functional improvement in subjects with chronic stroke.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of unilateral hemiparesis secondary to cerebrovascular accident with post-onset duration of more than 6 months
* ability to walk independently for at least 6 meters with or without use of walking aids
* ability to follow simple verbal commands or instructions

Exclusion Criteria:

* unstable medical conditions
* history of other diseases known to interfere with participation in the study
* past history of a seizure
* history of skin allergy to electrode
* use of a cardiac pacemaker

Ages: 40 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2008-08; Primary Completion 2008-12 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
N1 latency of somatosensory evoked potential | Change from baseline at 4 weeks
N1P1 amplitude of somatosensory evoked potential | Change from baseline at 4 weeks
motor threshold of motor evoked potential | Change from baseline at 4 weeks
map size of motor evoked potential | Change from baseline at 4 weeks

SECONDARY OUTCOMES:
Fugl-Meyer Assessment | Change from baseline at 4 weeks
Motricity Index | Change from baseline at 4 weeks
Berg Balance Scale | Change from baseline at 4 weeks
walking speed | Change from baseline at 4 weeks
Modified-Emory Functional Ambulation Profile | Change from baseline at 4 weeks
  Measures a patient's ability to walk through 5 commonly experienced types of terrain.